CLINICAL TRIAL: NCT07087626
Title: Prediction of Perioperative Complication Risk Using Chronic Obstructive Pulmonary Disease Assessment Test Score in Chronic Obstructive Pulmonary Disease Patients: A Prospective Cohort Study
Brief Title: COPD Assessment Test Score and Perioperative Risk in COPD
Acronym: COPD
Status: Not yet recruiting | Type: Observational
Sponsor: Erzurum City Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Sercan Orbak, Anesthesiology Specialist (MD), Erzurum City Hospital
Other Study IDs: ECH-AR-MSO-01
Record Dates: First submitted 2025-07-10; First posted 2025-07-28 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: COPD; Preoperative Risk Assessment
Keywords: COPD Assessment Test; COPD; Postoperative Respiratory Complications; Preoperative Risk Assessment
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Blood Gas Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CAT <10 (Low symptom burden): Patients scheduled for elective surgery, diagnosed with COPD in a stable stage according to the GOLD (Global Initiative for Chronic Obstructive Lung Disease) criteria, and identified as having a low symptom burden (CAT <10) based on preoperative CAT scoring
  Interventions: Other: Arterial Blood Gas Analysis
- CAT ≥10 (High symptom burden): Patients scheduled for elective surgery, diagnosed with COPD in a stable stage according to the GOLD (Global Initiative for Chronic Obstructive Lung Disease) criteria, and identified as having a high symptom burden (CAT ≥10) based on preoperative CAT scoring
  Interventions: Other: Arterial Blood Gas Analysis

INTERVENTIONS:
Other: Arterial Blood Gas Analysis — Arterial blood gas analysis will be performed at predefined time points: at rest during the preoperative period, before induction and preoxygenation during the perioperative period, two minutes after induction but prior to intubation, within the first 30 minutes in the PACU during the postoperative period, and at the 72nd postoperative hour in the ward

SUMMARY:
The goal of this observational cohort study is to evaluate whether the COPD Assessment Test (CAT) score can predict the risk of perioperative respiratory complications in patients aged 40 to 70 years with diagnosed Chronic Obstructive Pulmonary Disease (COPD), undergoing elective surgical procedures lasting no longer than 150 minutes.

The main questions it aims to answer are:

* Is there a statistically significant association between preoperative CAT scores and the incidence of intraoperative and early postoperative respiratory complications in COPD patients?
* Can the CAT score be effectively used as a preoperative risk stratification tool to guide anesthetic and surgical decision-making?

Researchers will compare two patient groups based on CAT scores: those with CAT <10 and those with CAT ≥10 to determine whether higher CAT scores are associated with an increased incidence of perioperative respiratory complications.

Participants will:

* Complete the CAT questionnaire during the preoperative evaluation
* Undergo elective surgery with an expected duration of ≤150 minutes
* Be monitored intraoperatively for bronchospasm, oxygen desaturation, and ventilation difficulty
* Be monitored postoperatively (within the first 72 hours) for hypoxemia, reintubation, bronchospasm episodes, postoperative pneumonia, intensive care unit (ICU) admission, and length of hospital stay
* Have perioperative clinical data collected and analyzed for comparative outcomes between CAT score subgroups

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a common chronic respiratory disease associated with increased perioperative morbidity and mortality. Surgical procedures in COPD patients often carry higher risks of respiratory complications, making anesthetic management more challenging. The COPD Assessment Test (CAT) is a simple and practical tool developed to assess symptom burden in COPD patients and is being increasingly integrated into clinical practice. While its utility in evaluating disease-related symptoms and quality of life is well documented, the role of CAT score in predicting perioperative respiratory complications remains unclear.

This prospective observational cohort study aims to evaluate whether the CAT score can be used to predict perioperative respiratory risk and support clinical decision-making for anesthesiology and surgical teams. Based on previous estimates, patients with high CAT scores appear to be at greater risk for complications. A total of 120 patients will be enrolled in the study, with 60 patients in each group. Patients will be categorized into two groups based on their CAT scores:

Group 1: CAT <10 (Low symptom burden)

Group 2: CAT ≥10 (High symptom burden)

Patients aged 40-70 years with a diagnosis of stable COPD scheduled for elective surgery lasting no more than 150 minutes will be included. The relationship between CAT score and perioperative respiratory complications will be statistically analyzed.

In the preoperative period (within 24 hours before surgery), data will be collected on demographics (age, sex, BMI, smoking history), comorbidities, surgical type (e.g., thoracic, abdominal, urological), ASA physical status classification, and planned anesthesia technique (general or regional). Arterial blood gas (ABG) samples at rest will be obtained. Additionally, Global Initiative for Chronic Obstructive Pulmonary Disease (GOLD) stage, spirometry data (Forced Expiratory Volume in 1 Second (FEV1), Forced Vital Capacity (FVC), FEV1/FVC ratio), and CAT score will be recorded by a pulmonologist.

During the perioperative period, ABG samples will be taken prior to induction and preoxygenation. All patients will receive standardized general anesthesia with full monitoring (Electrocardiogram (ECG), Peripheral Capillary Oxygen Saturation (SpO2), non-invasive blood pressure, capnography). Preoxygenation will be performed for at least 2 minutes. Anesthesia induction protocol includes:

* 1-2 mg IV midazolam (premedication)
* 0.3-0.5 mg/kg IV lidocaine
* 1.5-2.5 mg/kg IV propofol
* 0.6-1.2 mg/kg IV rocuronium
* 1-2 mcg/kg IV fentanyl

After sufficient muscle relaxation, endotracheal intubation will be performed. All patients will be ventilated using volume-controlled ventilation with ideal body weight-based settings: tidal volume 6-8 mL/kg, respiratory rate 10-14/min, Positive End-Expiratory Pressure (PEEP) 3-5 cmH₂O, I:E ratio 1:2, and target End-Tidal Carbon Dioxide (EtCO₂) of 35-45 mmHg. Volatile anesthetics (sevoflurane or desflurane) will be administered at a minimum of 1.3 Minimum Alveolar Concentration (MAC). Intraoperative respiratory events (bronchospasm, desaturation, ventilation difficulty) will be observed and documented. A second ABG sample will be collected 2 minutes after induction.

At the end of surgery, patients will receive 10-15 mg/kg IV paracetamol and 1-2 mg/kg IV tramadol for analgesia. Neuromuscular blockade will be reversed with 2 mg/kg IV sugammadex.

Postoperatively, ABG samples will be taken in the Post-Anesthesia Care Unit (PACU) and again at the 72nd hour. The following respiratory complications will be recorded within the first 72 hours:

* Hypoxemia (SpO₂ <92%)
* Reintubation requirement
* Bronchospasm episodes
* Postoperative pneumonia
* Intensive Care Unit (ICU) admission
* Length of hospital stay (in days)

All data will be collected by anesthesiologists involved in the study.

The primary objective of this study is to evaluate whether the preoperative CAT score can predict postoperative respiratory complications in patients with COPD. The secondary objective is to determine whether patients with high CAT scores require more postoperative oxygen therapy. The tertiary (exploratory) objective is to assess whether patients with higher CAT scores need more extensive medical optimization before surgery and whether the CAT score can serve as a useful guide in preoperative planning.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 40 and 70 years
* Diagnosed with stable-stage Chronic Obstructive Pulmonary Disease (COPD) according to GOLD criteria
* Scheduled for elective surgical intervention
* Classified as ASA Physical Status II or III according to the American Society of Anesthesiologists (ASA)
* Planned for postoperative follow-up and eligible for at least 72 hours of observation
* Undergoing surgery with an expected duration of at least 150 minutes
* Willing to participate voluntarily in the study

Exclusion Criteria:

* Patients younger than 40 years or older than 70 years
* History of COPD exacerbation within the past 4 weeks
* Presence of severe cardiac failure (EF <30%), end-stage renal disease, or active malignancy
* Neurological disorders or cognitive impairments
* Requirement for invasive mechanical ventilation in the preoperative period
* Altered consciousness or any condition preventing completion of forms before anesthesia
* Undergoing surgery with an expected duration longer than 150 minutes
* Unwillingness to participate in the study voluntarily

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged between 40 and 70 years with a diagnosis of stable-stage COPD according to GOLD criteria
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative Respiratory Complications Within 72 Hours | Within 72 hours postoperatively
  Respiratory complications including hypoxemia (SpO₂ < 90%), reintubation, bronchospasm, pneumonia, or ICU admission will be recorded during the first 72 hours after surgery. Each event will be assessed based on standardized clinical definitions.
  The outcome will be reported as the number of patients who experience at least one of the defined complications.

SECONDARY OUTCOMES:
Initiation of Postoperative Oxygen Therapy | Within 72 hours postoperatively
  The requirement for supplemental oxygen within 72 hours after surgery will be recorded. Supplemental oxygen therapy will be initiated based on predefined clinical criteria such as SpO₂ < 92% or signs of respiratory distress.
  The outcome will be reported as the number of patients who required oxygen therapy.
Duration of Postoperative Oxygen Therapy | Within 72 hours postoperatively
  The total duration of postoperative oxygen therapy will be recorded for each patient from initiation to discontinuation, within the first 72 hours after surgery. The outcome will be reported as the number of hours per patient receiving oxygen therapy.
Maximum Oxygen Flow Rate Administered Postoperatively | Within 72 hours postoperatively
  The highest flow rate of supplemental oxygen administered to each patient during the first 72 hours after surgery will be documented. The outcome will be expressed in liters per minute (L/min).

OTHER OUTCOMES:
Number of Patients Requiring Preoperative Medical Optimization | From preoperative assessment to day of surgery
  The total number of COPD patients requiring preoperative medical optimization interventions prior to surgery will be recorded. The outcome will be expressed as the number of patients who received such interventions, including respiratory therapy adjustments, medication changes, or pulmonology consultations.
Types of Preoperative Interventions Performed | From preoperative assessment to day of surgery
  A categorized record of preoperative medical interventions will be documented, including types such as bronchodilator adjustment, initiation of new medications, and pulmonology consultation. The outcome will be reported as the count of each intervention type (category-wise frequency).

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet S Orbak, Principal Investigator — Erzurum City Hospital
Locations (1):
- Erzurum City Hospital, Erzurum, Yakutiye, Turkey (Türkiye)